CLINICAL TRIAL: NCT01230307
Title: D suppLementation In HearT FaiLure (DELIGHTFUL)
Brief Title: Vitamin D Supplementation for Treatment of Heart Failure
Acronym: DELIGHTFUL
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit sufficient number of patients.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Barry E. Bleske, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VitD3
Record Dates: First submitted 2010-10-27; First posted 2010-10-29 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-09

CONDITIONS: Heart Failure
Keywords: Vitamin D; Systolic failure; Genomics; Biomarkers; Exercise; Quality of Life
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Cholecalciferol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Active Comparator): Vitamin D supplementation will be an oral load of 100,000 IU then 2000 IU by mouth daily of vitamin D3 (cholecalciferol)for 6 months
  Interventions: Drug: Vitamin D3
- Placebo (Placebo Comparator): A placebo loading dose will be given followed by two placebo tablets daily for 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D supplementation will be an oral load of 100,000 IU then 2000 IU by mouth daily of vitamin D3 (cholecalciferol)for 6 months
  Other Names: cholecalciferol
  Arms: Vitamin D
Drug: Placebo — A placebo loading dose will be given followed by 2 placebo tablets daily for 6 months.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The central objective of this proposal is to establish that vitamin D supplementation in heart failure patients with low vitamin D levels will have improved outcomes compared to placebo. In addition the investigators will also evaluate the role of genetics in regard to vitamin D and heart failure. The investigators will be evaluating what is currently a novel approach of identifying patients with low vitamin D and treating this low vitamin D level. The investigators will be able to evaluate the importance of vitamin D supplementation in these patients and the role of genetics on our defined outcomes.

DETAILED DESCRIPTION:
Primary Objective To determine how rapid vitamin D supplementation affects biomarkers and submaximal exercise capacity in systolic HF patients with low vitamin D status.

Working Hypothesis 1: HF patients when supplemented with vitamin D for 6 months will have lower measures of inflammation and extracellular-matrix remodeling compared with placebo.

Working Hypothesis 2: HF patients when supplemented with vitamin D for 6 months will have longer 6-minute walk length compared with placebo.

Secondary Objectives To establish a relationship between the CYP2R1 variant and surrogate markers in systolic HF patients.

Working Hypothesis 3: HF patients with the CYP2R1 G allele will have higher measures of inflammation and extracellular-matrix remodeling compared to AA subjects. This relationship will also be seen in subjects with the CYP2R1 TagSNP variants.

Working Hypothesis 4: HF patients with CYP2R1 variant alleles will have shorter 6-minute walk length compared to subjects without these variants.

To genotype HF subjects for the VDR variants and additional tag SNPs, to ascertain the relationship between VDR genetic variation and surrogate markers in systolic HF patients.

Working Hypothesis 5: HF patients with VDR variants will have greater measures of inflammation and extracellular-matrix remodeling compared to subjects without VDR variants.

Working Hypothesis 6: HF patients with VDR variants will have a shorter 6-minute walk length compared to subjects without these variants.

ELIGIBILITY:
Inclusion Criteria:

* HF patients with LV systolic dysfunction of ischemic or non-ischemic origin and an LVEF <40% using nuclear ventriculography or echocardiography within the last 6 months.
* Attempts should have been made at optimizing medical therapy and the participant should be stable on these medications for at least 3 months.
* Patients with a 25(OH)D level between 10-25 ng/ml

Exclusion Criteria:

* Inability to give informed consent
* Patients with sarcoidosis or other granulomatous disease that can alter vitamin D metabolism
* Patients with primary valvular HF, hypertrophic cardiomyopathy, and drug-induced HF
* Renal dysfunction defined as serum creatinine > 2.5 mg/dl
* Pregnant women
* Patients <18 years of age
* Patients on vitamin D supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry E. Bleske, Pharm. D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Medical Center, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16 consented participants were not randomized due to screen fails.
Period: Overall Study
Arm/Group | Vitamin D | Placebo
Started | 6 | 6
Completed | 6 | 4
Not Completed | 0 | 2
Not completed — LVAD Placement | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Customized [Number; unit: participants]
  46 - 78 Years | 6 | 6 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 6 | 4 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 5 | 5 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Baseline Vit D level (ng/mL) [Mean (Standard Deviation); unit: ng/mL] — Baseline Vit D level nanograms per milliliter of blood.
  ng/mL | 16.3 (5) | 19.6 (3) | 17.8 (4)

OUTCOME MEASURES:

1. Primary Outcome: Biomarkers
Description: Biomarkers - C-reactive protein (CRP), interleukin-6 (IL-6), tumor necrosis factor-a (TNF-a), propeptide procollagen type I, plasma procollagen III, matrix metalloproteinase 2 (MMP-2), MMP-9 and tissue inhibitor of matrix metalloproteinases-1 (TIMP-1).
Time Frame: 6 months
Population: Because enrollment was less than 30% of original goal (6 vs 4 subjects) and therefore would not have scientific validity and would be a waste of financial resources, this outcome was not analyzed.
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Exercise Capacity Measured by 6 Minute Walk Test
Time Frame: 6 months
Population: Because enrollment was less than 30% of original goal (6 vs 4 patients) and therefore would not have scientific validity and no conclusions could be determined, this outcome was not analyzed.
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quality of Life Measured by Kansas City Cardiomyopathy Questionnaire
Description: Kansas City Cardiomyopathy Questionnaire for quality of life is measured on a scale of 0 - 100, with 100 being best.
Time Frame: 6 months
Population: as for outcome 2
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Vitamin D Genomics
Description: Genotyped for the restricted fragment length polymorphism at the BsmI site. In addition CYP2R1, CYP27B1, CYP24 will also be genotyped.
Time Frame: Baseline
Population: Because enrollment was less than 30% of original goal (6 vs 4 patients) and therefore would not have scientific validity, in addition there is significant time and costs associated with this measurement which would result in data that would lead to no conclusions, this outcome was not analyzed.
Arm/Group | Vitamin D | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vitamin D | Placebo
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D (N=6) | Placebo (N=6)
GI bleed (Gastrointestinal disorders) | 1 (1) | 0 (0)
syncope due to hypokalemia (Nervous system disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Only a fraction of the original goal of enrollment was met. Therefore, analysis of comparative results was not done. No conclusions of any kind can be made from analyzing the data with the number of patients completing the trial (6 vs 4 patients).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No